CLINICAL TRIAL: NCT05464004
Title: Effects of Nintendo Wii Balance Board in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0706
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Balance Problem; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Effects of Nintendo Wii balance board in combination with conventional physical therapy in children with CP
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy (Active Comparator): stretching, strengthening and balance exercises
  Interventions: Other: Nintendo Wii balance board
- Nintendo Wii balance board therapy (Experimental): Nintendo Wii balance board therapy in combination with conventional physical therapy
  Interventions: Other: Nintendo Wii balance board

INTERVENTIONS:
Other: Nintendo Wii balance board — Experimental group was given Nintendo Wii balance board therapy in combination with conventional physical therapy for 16 sessions/8 weeks
  Control group was conventional physical therapy which include stretching of the hamstrings, quadriceps and calf muscles. strengthening of the lower limb. Balance exercises include walk in parallel bar
  Other Names: Conventional physical therapy

SUMMARY:
I wan to check the effects of Nintendo Wii balance board therapy in children with CP.

DETAILED DESCRIPTION:
Evaluate the effects of Nintendo Wii balance board therapy in combination with conventional physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* children with age of 7-14 years. No history of falls. children able to stand independently. delays in gait development.

Exclusion Criteria:

* Children with hemiplegic CP. Comorbidities. children with lower limb contractures. hearing disorders. children with epilepsy.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Effects of Nintendo Wii balance board in children with CP | 8th week
  Changes from the baseline. it was designed to measure the balance issues in children with pediatric balance scale and pediatric forward reach test. it consist of 14 items and total score of 56

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, MS, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Gage JR, Novacheck TF. An update on the treatment of gait problems in cerebral palsy. J Pediatr Orthop B. 2001 Oct;10(4):265-74. PMID 11727367
- [Background] Woollacott MH, Shumway-Cook A. Postural dysfunction during standing and walking in children with cerebral palsy: what are the underlying problems and what new therapies might improve balance? Neural Plast. 2005;12(2-3):211-9; discussion 263-72. doi: 10.1155/NP.2005.211. PMID 16097489
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598